CLINICAL TRIAL: NCT03549988
Title: Pro-active Fecal Calprotectin Monitoring to Improve Patient Outcomes in Ulcerative Colitis: A Prospective Randomised Control Trial
Brief Title: Pro-active Fecal Calprotectin Monitoring PROMOTE-UC
Status: Active, not recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Greg Rosenfeld, Clinical Assistant Professor, University of British Columbia
Other Study IDs: H18-00647
Record Dates: First submitted 2018-05-05; First posted 2018-06-08 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Fecal calprotectin
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: The group will receive current standard of care as the usual practice of the attending physician. Basic research data will be collected and participants in this group will be asked to complete the on-line questionnaires (SIBDQ and EQ-5D 5L) on the baseline visit and month 6, 12 and month 18.
  When endoscopy is performed biopsies should be taken and the endoscopic and histologic assessment will be recorded. If a fecal calprotectin is measured, every effort should be made to use the IBDoc with the result being sent to the central primary investigator via the IBDoc Web Portal. However, should a different fecal calprotectin measure be used, this will be recorded as part of the study documentation and will be included in the study data.
- Intervention: FC measurements with IBDoc: Fecal Calprotectin (FC) measurements with IBDocTM home kits will be performed by participants in the intervention group every 2 months until final visit.
  Basic research data will be collected and participants in this group will be asked to complete the on-line questionnaires (SIBDQ and EQ-5D 5L) on baseline visit and month 6, 12 and month 18.
  Interventions: Other: Fecal Calprotectin (FC) measurements with IBDocTM

INTERVENTIONS:
Other: Fecal Calprotectin (FC) measurements with IBDocTM — Each IBDocTM kit measure one fecal calprotectin value. The IBDoc® is an in-vitro diagnostic immunoassay analyzed by a downloadable smartphone application (CalApp®). A patient is able to process their stool at home using a test cassette.
  The IBDocTM test results are displayed in a light signal system as three titre categories; normal <100 µg/g (green), 100-300 µg/g (yellow), >300 µg/g (high). Patients' results will be sent directly to the central research coordinator through the IBDoc® Web Portal. If the FC is >250 µg/g a second FC will be performed within 2 weeks. If this result is <250 µg/g patients will continue to monitor their FC every 2 months. If the second result is >250 µg/g, the attending physician will review the patient either by telephone or in the office within 7 days.
  Groups: Intervention: FC measurements with IBDoc

SUMMARY:
Hypothesis:

Pro-active home fecal calprotectin testing in patients with Ulcerative Colitis will allow early detection and treatment of inflammation to prevent symptomatic flares. This will result in less steroid use, fewer hospitalizations and a reduced risk of surgery, as well as improved quality of life and adherence to medication.

DETAILED DESCRIPTION:
Previous studies have shown that fecal calprotectin (FC) may be useful to predict relapse of inflammatory bowel disease and response to treatment. Current methods for measurement of FC require bringing stool samples to the laboratory or physician's office. The test is either not readily available or is expensive for patients. Some patients also find it inconvenient to collect, transport and travel to return the sample.

A prior study in our institution showed that only 77% of patients returned samples for processing. Therefore, a home-based kit may offer greater uptake by patients as samples do not need to be returned to a lab or physician's office. Regular monitoring of patients at home may allow the detection and prediction of flares before the appearance of symptoms. With earlier treatment, the risk of complications may be minimized and the quality of life for people living with this disease may be improved.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 19 years or older with Ulcerative Colitis
* Symptomatic remission defined as a modified Partial Mayo score ≤ 2 with a rectal bleeding score = 0
* Able to use IBDocTM test kit which requires a smart phone with a camera and internet access to download the CalApp® which interprets the measurement
* Able to give informed consent to the study protocol

Exclusion Criteria:

* Patients experiencing a symptomatic flare
* Patients currently receiving therapy as part of a clinical trial
* Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of 756 patients with Ulcerative colitis in symptomatic remission. Through the Canadian Intestinal Research Consortium (CIRC), we intent to involve a minimum of 12 sites across Canada, Europe and Australia.
Sampling Method: Probability Sample
Enrollment: 726 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The time to a symptomatic flare, defined as an increase in modified partial Mayo score > 2 points from baseline or a rectal bleeding score > 1 | 6 months
  All patients in both control and intervention group will be contacted every 6 months until end of study. Partial Mayo and rectal bleeding score will be obtained and if there is an increase in partial Mayo score > 2 points from baseline or a rectal bleeding score > 1, this is considered as flare. Endoscopy will be performed wherever possible.

SECONDARY OUTCOMES:
Hospitalization, surgery, steroid or biologic use | 6 months
  All patients in both control and intervention group will be asked every 6 months whether they were hospitalized, had undergone surgery, had used steroid (oral or rectal) or any biologics.
Proportion of subjects who underwent an escalation of therapy | 6 months
  Choice of therapy for all patients should be according to the standard of care and by the judgement of the attending physician.
Quality of life measured by SIBDQ questionnaire | 6 months
  Quality of life is measured by Short Quality of Life in Inflammatory Bowel Disease (SIBDQ) questionnaire. Both control and intervention group will be asked to complete these questionnaires on-line during baseline, month 6, 12 and month 18.
  The SIBDQ provide a measure of subjective health status or quality of life in patients with inflammatory bowel disease (IBD). It consists of four domains, bowel symptoms, emotional health, systemic systems and social function. The total score ranges from 10 (worst health) to 70 (best health).
Quality of life measured by EQ-5D 5L questionnaire | 6 months
  Quality of life is measured by EQ-5D 5L health questionnaire. Both control and intervention group will be asked to complete these questionnaires on-line during baseline, month 6, 12 and month 18.
  The EQ-5D-5L is a standardized measure of health status. It comprises of 5 dimensions like mobility, selfcare, usual activities, pain/discomfort, anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The patient is asked to indicate his/her health state. This decision results in a 1-digit number expressing the level selected for that dimension. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state.
Number of physician visits | 6 months
  Participants will be asked the number of physician visits during the course of the study.
Time lost from work or school | 6 months
  Participants will be asked about time lost from work or school because of ulcerative colitis symptoms.
Correlation of fecal calprotectin with endoscopic activity | 6 months
  Endoscopic disease activity is measured by Mayo score. The Mayo Endoscopic Score is classified into the following four categories: 0, normal mucosa or inactive disease; 1, mild disease with erythema, decreased vascular patterns and mild friability; 2, moderate disease with marked erythema, absence of vascular patterns, friability and erosions; 3, severe disease with spontaneous bleeding and ulceration.
Correlation of fecal calprotectin with histologic disease activity | 6 months
  A histologic scoring index is a system used to assess the patient's disease severity using tissue sample. In this study, the Robarts Histology Index (RHI) is used. The RHI can be calculated as 1 x chronic inflammatory infiltrate (4 levels) plus 2 x lamina propria neutrophils (4 levels) plus 3 x neutrophils in epithelium (4 levels) plus 5 x erosion or ulceration (4 levels after combining Geboes 5:1 and 5:2).
  Score takes into consideration histologic variables like crypt abscesses, presence of granulation tissue or aggregates of inflammatory elements in the superficial part of the mucosa, indicative of erosions or ulcers, neutrophils in the lamina propria.
Successful use of IBDoc | 2 months
  Successful use of IBDoc home test kits will be measured by the completed test reported in the IBDoc portal.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Rosenfeld, MD, Principal Investigator — University of British Columbia, Depart. of Medicine, Div. of Gastroenterology
Locations (1):
- Pacific Gastroenterology Associates, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Bernstein CN, Wajda A, Svenson LW, MacKenzie A, Koehoorn M, Jackson M, Fedorak R, Israel D, Blanchard JF. The epidemiology of inflammatory bowel disease in Canada: a population-based study. Am J Gastroenterol. 2006 Jul;101(7):1559-68. doi: 10.1111/j.1572-0241.2006.00603.x. PMID 16863561
- [Background] Rocchi A, Benchimol EI, Bernstein CN, Bitton A, Feagan B, Panaccione R, Glasgow KW, Fernandes A, Ghosh S. Inflammatory bowel disease: a Canadian burden of illness review. Can J Gastroenterol. 2012 Nov;26(11):811-7. doi: 10.1155/2012/984575. PMID 23166905
- [Background] Roseth AG, Aadland E, Jahnsen J, Raknerud N. Assessment of disease activity in ulcerative colitis by faecal calprotectin, a novel granulocyte marker protein. Digestion. 1997;58(2):176-80. doi: 10.1159/000201441. PMID 9144308
- [Background] Costa F, Mumolo MG, Ceccarelli L, Bellini M, Romano MR, Sterpi C, Ricchiuti A, Marchi S, Bottai M. Calprotectin is a stronger predictive marker of relapse in ulcerative colitis than in Crohn's disease. Gut. 2005 Mar;54(3):364-8. doi: 10.1136/gut.2004.043406. PMID 15710984
- [Background] Kopylov U, Rosenfeld G, Bressler B, Seidman E. Clinical utility of fecal biomarkers for the diagnosis and management of inflammatory bowel disease. Inflamm Bowel Dis. 2014 Apr;20(4):742-56. doi: 10.1097/01.MIB.0000442681.85545.31. PMID 24562174
- [Background] Zhulina Y, Cao Y, Amcoff K, Carlson M, Tysk C, Halfvarson J. The prognostic significance of faecal calprotectin in patients with inactive inflammatory bowel disease. Aliment Pharmacol Ther. 2016 Sep;44(5):495-504. doi: 10.1111/apt.13731. Epub 2016 Jul 12. PMID 27402063
- [Background] Rosenfeld G, Greenup AJ, Round A, Takach O, Halparin L, Saadeddin A, Ho JK, Lee T, Enns R, Bressler B. FOCUS: Future of fecal calprotectin utility study in inflammatory bowel disease. World J Gastroenterol. 2016 Sep 28;22(36):8211-8. doi: 10.3748/wjg.v22.i36.8211. PMID 27688663
- [Background] Trindade AJ, Ehrlich A, Kornbluth A, Ullman TA. Are your patients taking their medicine? Validation of a new adherence scale in patients with inflammatory bowel disease and comparison with physician perception of adherence. Inflamm Bowel Dis. 2011 Feb;17(2):599-604. doi: 10.1002/ibd.21310. PMID 20848512
- [Background] Jowett SL, Seal CJ, Barton JR, Welfare MR. The short inflammatory bowel disease questionnaire is reliable and responsive to clinically important change in ulcerative colitis. Am J Gastroenterol. 2001 Oct;96(10):2921-8. doi: 10.1111/j.1572-0241.2001.04682.x. PMID 11693327
- [Background] Agborsangaya CB, Lahtinen M, Cooke T, Johnson JA. Comparing the EQ-5D 3L and 5L: measurement properties and association with chronic conditions and multimorbidity in the general population. Health Qual Life Outcomes. 2014 May 16;12:74. doi: 10.1186/1477-7525-12-74. PMID 24885017
- [Background] Mosli MH, Feagan BG, Zou G, Sandborn WJ, D'Haens G, Khanna R, Shackelton LM, Walker CW, Nelson S, Vandervoort MK, Frisbie V, Samaan MA, Jairath V, Driman DK, Geboes K, Valasek MA, Pai RK, Lauwers GY, Riddell R, Stitt LW, Levesque BG. Development and validation of a histological index for UC. Gut. 2017 Jan;66(1):50-58. doi: 10.1136/gutjnl-2015-310393. Epub 2015 Oct 16. PMID 26475633
- [Background] Bressler B, Marshall JK, Bernstein CN, Bitton A, Jones J, Leontiadis GI, Panaccione R, Steinhart AH, Tse F, Feagan B; Toronto Ulcerative Colitis Consensus Group. Clinical practice guidelines for the medical management of nonhospitalized ulcerative colitis: the Toronto consensus. Gastroenterology. 2015 May;148(5):1035-1058.e3. doi: 10.1053/j.gastro.2015.03.001. Epub 2015 Mar 4. PMID 25747596
- [Background] Heida A, Knol M, Kobold AM, Bootsman J, Dijkstra G, van Rheenen PF. Agreement Between Home-Based Measurement of Stool Calprotectin and ELISA Results for Monitoring Inflammatory Bowel Disease Activity. Clin Gastroenterol Hepatol. 2017 Nov;15(11):1742-1749.e2. doi: 10.1016/j.cgh.2017.06.007. Epub 2017 Jun 10. PMID 28606846
- [Background] Bello C, Roseth A, Guardiola J, Reenaers C, Ruiz-Cerulla A, Van Kemseke C, Arajol C, Reinhard C, Seidel L, Louis E. Usability of a home-based test for the measurement of fecal calprotectin in asymptomatic IBD patients. Dig Liver Dis. 2017 Sep;49(9):991-996. doi: 10.1016/j.dld.2017.05.009. Epub 2017 May 19. PMID 28587751
- [Background] Feagan BG, Macdonald JK. Oral 5-aminosalicylic acid for induction of remission in ulcerative colitis. Cochrane Database Syst Rev. 2012 Oct 17;10:CD000543. doi: 10.1002/14651858.CD000543.pub3. PMID 23076889